CLINICAL TRIAL: NCT05690477
Title: Corrective Osteotomy of the Distal Radius With Palmar Locking Plate Osteosynthesis Without Bone Grafting and Without Cortical Contact
Brief Title: Corrective Osteotomy of the Distal Radius Without Bone Grafting
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Vilijam Zdravkovic, Dr. med., Cantonal Hospital of St. Gallen
Other Study IDs: 27012022
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Corrective osteotomy of the distal radius — Corrective osteotomy of the distal radius with a palmar locking plate osteosynthesis without the use of a bone graft and without cortical contact.

SUMMARY:
The investigators retrospectively analyzed patients who underwent extraarticular corrective osteotomy of the distal radius via a palmar approach and without the use of a bone graft, even in the absence of cortical contact after corrective osteotomy.

The goal of this retrospective observational study is to determine whether secondary dislocation or nonunion occurs after corrective osteotomy without bone grafting.

ELIGIBILITY:
Inclusion Criteria:

* malunited distal radius fracture
* extraarticular corrective osteotomy
* palmar approach
* no bone graft used
* no cortical contact after dorsal open wedge osteotomy
* signed informed consent

Exclusion Criteria:

* others reasons for malunion
* intraarticular corrective osteotomy
* use of a bone graft
* cortical contact after open wedge osteotomy
* lost to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with extraarticular corrective osteotomy of the distal radius without cortical contact and without the use of bone graft due to a malunited distal radius fracture
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Secondary fracture dislocation | 1 year
complete bone healing | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hand, Plastic and Reconstructive Surgery, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuchs J, Spuhler DL, Luz S, Zdravkovic V, Hainich J. Corrective osteotomy of the distal radius with palmar locking plate osteosynthesis without bone grafting and without cortical contact. J Hand Surg Eur Vol. 2024 Mar;49(3):359-365. doi: 10.1177/17531934231179875. Epub 2023 Jun 13. PMID 37310077